CLINICAL TRIAL: NCT02581787
Title: Fresolimumab and Stereotactic Ablative Radiotherapy in Early Stage Non-small Cell Lung Cancer
Brief Title: SABR-ATAC: A Trial of TGF-beta Inhibition and Stereotactic Ablative Radiotherapy for Early Stage Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maximilian Diehn (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor-Investigator, Maximilian Diehn, Assistant Professor of Radiation Oncology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-34863; NCI-2015-01726 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LUN0071 (Other: Stanford Cancer Institute); IRB-34863 (Other: Stanford IRB)
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Stage IA Non-Small Cell Lung Carcinoma; Stage IB Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — fresolimumab; Immunoglobulin G; Disulfides; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- (Phase 1) Fresolimumab 3 mg/kg (Experimental): Patients receive fresolimumab 3 mg/kg IV on days 1, 15, and 36 and undergo SABR in 4 fractions between days 8 and 12.
  Interventions: Biological: Fresolimumab; Radiation: Stereotactic Body Radiation Therapy
- (Phase 1) Fresolimumab 1 mg/kg (Experimental): Patients receive fresolimumab 1 mg/kg IV on days 1, 15, and 36 and undergo SABR in 4 fractions between days 8 and 12.
  Interventions: Biological: Fresolimumab; Radiation: Stereotactic Body Radiation Therapy
- (Phase 2) Fresolimumab (Experimental): Fresolimumab will be administered IV at the dose selected in the preceding Phase 1 on Days 1, 15 and 36 and SABR will be administered in 4 fractions between Days 8 and 12.
  Interventions: Biological: Fresolimumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Biological: Fresolimumab — Given IV
  Other Names: Anti-TGF-Beta Monoclonal Antibody GC1008; GC1008; Human Anti-TGF-Beta Monoclonal Antibody GC1008; Immunoglobulin G4, anti-(transforming growth factor beta) (human monoclonal GC-1008 heavy chain), disulfide with human monoclonal GC-1008 light chain, Dimer
Radiation: Stereotactic Body Radiation Therapy — Undergo SABR
  Other Names: SBRT

SUMMARY:
The SABR-ATAC trial (Stereotactic Ablative Radiotherapy and anti-TGFB Antibody Combination) is a phase I/II trial that studies the side effects and efficacy of fresolimumab, an anti-transforming growth factor beta (TGFB) antibody, when given with stereotactic ablative radiotherapy in patients with stage IA-IB non-small cell lung cancer. Fresolimumab may inhibit radiation side effects and block tumor growth through multiple mechanisms. Stereotactic ablative radiotherapy (SABR), also known as stereotactic body radiotherapy (SBRT), is a specialized form of radiation therapy that precisely delivers high dose radiation directly to tumors, thus killing tumor cells and minimizing damage to normal tissue. Giving fresolimumab with SABR may work better in treating patients with early stage non-small cell lung cancer than treating with SABR alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Phase 1: Evaluate the safe dose of fresolimumab in combination with stereotactic ablative radiotherapy (SABR) in patients.

Phase 2. Evaluate the rate of radiation induced pulmonary fibrosis after SABR plus fresolimumab.

SECONDARY OBJECTIVES:

I. Evaluate potential adverse events in patients receiving fresolimumab plus SABR. (Phase I) II. Evaluate post treatment changes in pulmonary function. (Phase I) III. Evaluate recurrence rates and progression free survival. (Phase I) IV. Assess pharmacokinetics (PK) of fresolimumab in combination with SABR (optional for patient). (Phase I) V. Evaluate the rate and severity of radiation induced pulmonary fibrosis after SABR plus fresolimumab. (Phase I) VI. Evaluate the severity of radiation induced pulmonary fibrosis after SABR plus fresolimumab. (Phase II) VII. Evaluate potential adverse events in patients receiving fresolimumab plus SABR. (Phase II) VIII. Evaluate post treatment changes in pulmonary function. (Phase II) IX. Evaluate recurrence rates and progression free survival. (Phase II)

OUTLINE: This is a phase I, dose escalation study of fresolimumab followed by a phase II study.

* Phase 1: A cohort of 5 patients receive the pre-selected dose of 3mg/kg of fresolimumab. If one patient experiences a DLT, an additional 5 patients will be enrolled at 3 mg/kg. If no more patients experience a DLT, then 3 mg/kg will be the dose for the Phase 2 component. If 2 or more patients experience a DLT in the total expanded cohort (or 2 or more patients in the initial cohort experience DLT), then the investigational dose of fresolimumab will be changed to 1 mg/kg. If 2 or more patients in the initial cohort experience DLT before all 5 patients have been enrolled, the remaining patients will receive the lower dose of 1 mg/kg.
* Phase 2: Patients receive fresolimumab intravenously (IV) on days 1, 15, and 36 and undergo SABR in 4 fractions between days 8 and 12.

After completion of study treatment, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically proven (or strongly suspected, see below) T1-T2aN0M0 (Stage IA-IB) non-small cell lung cancer (NSCLC), with maximum tumor diameter =< 5 cm under consideration for stereotactic ablative body radiotherapy (SABR) as definitive primary treatment
* Patient judged to be inoperable or at high surgical risk by a board qualified thoracic cancer surgeon who has evaluated the subject within the prior 12 weeks, or the patient's case has been discussed at a multidisciplinary tumor board with a thoracic cancer surgeon in attendance, or a patient who refuses surgery or declines to be evaluated for surgery.
* Able to give informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2
* Men or women of child bearing potential must agree to use an acceptable method of birth control (hormonal or barrier method of birth control; abstinence) to avoid pregnancy for at least 90 days after last study treatment (radiation or fresolimumab)

Exclusion Criteria:

* Significant anemia (hemoglobin below 9.0 g/dL) or neutropenia (absolute neutrophil count [ANC] < 1000/mm^3)
* Prior history of multifocal adenocarcinoma in situ (ie, classic or pure bronchioloalveolar carcinoma)
* Prior history of keratoacanthoma (well differentiated squamous cell skin cancer variant, often centrally ulcerated); history of basal cell cancer is allowed
* Pre malignant skin lesion(s) noted on prescreening skin exam, except for actinic (solar) keratosis
* Prior radiotherapy overlapping with high dose region of planned SABR course
* Prior history of head and neck; oral; or bladder cancer
* Prior receipt of systemic treatment (chemotherapy, targeted therapy, or immunotherapy) for the lesion under consideration of treatment
* Uncontrolled, inter current or recent illness that in the investigator's opinion precludes participation in the study, including those undergoing therapy for a separate invasive malignancy
* Contraindication to receiving radiotherapy
* Known allergy to components of fresolimumab
* Pregnant or breastfeeding. All women of child bearing potential (last menstrual period within the previous 12 months and not surgically sterile) will be tested for pregnancy at pre entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Diehn, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 participants signed consent; 24 were allocated to treatment.
Period: Phase 1
Arm/Group | (Phase 1) Fresolimumab 3 mg/kg | (Phase 1) Fresolimumab 1 mg/kg | (Phase 2) Fresolimumab
Started | 5 | 0 | 0
Received Treatment | 5 | 0 | 0
Completed Radiation | 4 | 0 | 0
Completed FRESO Treatments | 4 | 0 | 0
Completed 12-month Follow-up Visit | 5 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 1 | 0 | 0
Period: Phase 2
Arm/Group | (Phase 1) Fresolimumab 3 mg/kg | (Phase 1) Fresolimumab 1 mg/kg | (Phase 2) Fresolimumab
Started | 0 | 0 | 19
Received Treatment | 0 | 0 | 18
Completed Radiation | 0 | 0 | 17
Completed FRESO Treatments | 0 | 0 | 13
Completed 12-month Follow-up Visit | 0 | 0 | 13
Completed | 0 | 0 | 12
Not Completed | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (Phase 1) Fresolimumab 3 mg/kg | (Phase 2) Fresolimumab | Total
Number analyzed (Participants) | 5 | 19 | 24
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 0 | 1 | 1
  60-69 years | 2 | 4 | 6
  70-79 years | 3 | 9 | 12
  80-89 years | 0 | 5 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 2 | 11 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 19 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 2 | 2
  White | 5 | 14 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 19 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicities (DLTs) of Fresolimumab When Combined With SABR (Phase I)
Description: DLT is defined as CTCAE grade 3 or higher radiation pneumonitis or bronchopulmonary hemorrhage.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | (Phase 1) Fresolimumab 3 mg/kg
Number analyzed (Participants) | 5
Participants | 0

2. Primary Outcome: Number of Participants With Late Radiation Induced Fibrosis
Description: Presence of radiation induced pulmonary fibrosis is defined as presence of a moderate-to-severe level of fibrosis. This outcome is primary in phase 2 patients.
Time Frame: 12 months
Population: Patients who met criteria to be considered for endpoint analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | (Phase 2) Fresolimumab
Number analyzed (Participants) | 15
Participants | 5

3. Secondary Outcome: Number of Participants With Late Radiation Induced Fibrosis (Phase 1 Patients)
Description: Presence of radiation induced pulmonary fibrosis is defined as presence of a moderate-to-severe level of fibrosis. This outcome is secondary for phase 1 patients.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | (Phase 1) Fresolimumab 3 mg/kg
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | (Phase 1) Fresolimumab 3 mg/kg | (Phase 2) Fresolimumab
All-Cause Mortality (participants affected / at risk) | 4/5 | 5/19
Serious Adverse Events (participants affected / at risk) | 0/5 | 6/19
Other Adverse Events (participants affected / at risk) | 5/5 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (Phase 1) Fresolimumab 3 mg/kg (N=5) | (Phase 2) Fresolimumab (N=19)
anemia (Blood and lymphatic system disorders) | 0 | 2
av block (Cardiac disorders) | 0 | 1
upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
lung infection (Infections and infestations) | 0 | 1
sepsis (Infections and infestations) | 0 | 1
dehydration (Metabolism and nutrition disorders) | 0 | 1
encephalopathy (Nervous system disorders) | 0 | 1
mental changes status (Nervous system disorders) | 0 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (Phase 1) Fresolimumab 3 mg/kg (N=5) | (Phase 2) Fresolimumab (N=19)
anemia (Blood and lymphatic system disorders) | 0 | 5
atrial fibrillation (Cardiac disorders) | 0 | 1
chest pain - cardiac (Cardiac disorders) | 0 | 1
esophagitis (Gastrointestinal disorders) | 0 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 1
bloating (Gastrointestinal disorders) | 0 | 1
dysphagia (Gastrointestinal disorders) | 0 | 1
mucositis oral (Gastrointestinal disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 2 | 1
edema limbs (General disorders) | 0 | 3
fatigue (General disorders) | 2 | 6
infusion related reaction (General disorders) | 0 | 1
non-cardiac chest pain (General disorders) | 0 | 1
r cheek skin lesion (Infections and infestations) | 0 | 1
upper respiratory infection (Infections and infestations) | 0 | 1
rash pustular (Infections and infestations) | 0 | 1
dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 3
creatinine increased (Investigations) | 0 | 2
weight loss (Investigations) | 0 | 2
lymphocyte count decreased (Investigations) | 0 | 1
wbc decreased (Investigations) | 0 | 1
lymphocyte count decrease (Investigations) | 0 | 1
anorexia (Metabolism and nutrition disorders) | 1 | 2
hyponatremia (Metabolism and nutrition disorders) | 0 | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 8
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
headache (Nervous system disorders) | 0 | 4
dizziness (Nervous system disorders) | 0 | 1
presyncope (Nervous system disorders) | 0 | 1
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
bronchial obstruction (copd) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1
hypertension (Vascular disorders) | 0 | 1
hypotension (Vascular disorders) | 0 | 1
papulopustular rash (Infections and infestations) | 1 | 0
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT02581787/Prot_SAP_001.pdf